CLINICAL TRIAL: NCT03966092
Title: Analgesic Effect of Bilateral Quadratus Lumborum Block in the End of Colorectal Laparosopic Surgery: a Prospective Randomized Pilot Study
Brief Title: Analgesic Effect of Bilateral Quadratus Lumborum Block in the End of Colorectal Laparosopic Surgery.
Acronym: Coloqual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2018 VIGNAUD_Coloqual; 2019-000277-23 (Other: ANSM)
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Post Operative Pain; Laparoscopic Colorectal Surgery
Keywords: Prospective randomized pilot study; Quadratus lumborum block; Quo R 40 score; Post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomization in 2 groups
  * Control group (usual practice): patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen and morphine. Antimicrobial prophylaxis is performed according to recommendations.
  * Experimental group: patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen and morphine. Antimicrobial prophylaxis is performed according to recommendations. In this group, a bilateral quadratus lumborum block, using 20 ml of ropivacaine 3, 75 mg/ml is performed at the end of surgery, using ultrasound guidance.
Who Masked: Participant
Masking Description: During the assess period, the participant and the research staff involved in the data collection will be blinded to the randomization group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual practice (No Intervention): Patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen and morphine. Antimicrobial prophylaxis is performed according to recommendations
- QLB block (Experimental): Patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen and morphine. Antimicrobial prophylaxis is performed according to recommendations.
  In addition, patients receiving a bilateral QLB at the end of the surgery
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Quadratus lumborum block — * Bilateral Quatratus lumborum block is performed with ultra sound guidance. The high frequency probe is placed right to the umbilicus, and slips laterally to the side to block. It allows showing the three belts of larges muscles of abdomen (External Oblicum, internal oblicum, and transversal of the abdomen). Laterally, these three are merging to from fascia transversalis. Under fascia transversalis, we can see quadratus lumborum muscle. Punction point in lateral, 1cm in the plan separating quadratus lumborum block and fascia transversalis
  * 20 ml of ropivacaïne 3.75mg/ml are injected after aspiration test. If in doubt, hydro localisation car be realised.
  Arms: QLB block

SUMMARY:
The primary purpose of COLOQUAL study is to demonstrate the superiority of analgesic effect of a bilateral quadratus lumborum block (QLB), performed at the end of laparoscopic colorectal surgery, compared to standard of care.

The investigators hypothesized that a bilateral quadratus lumborum block performed at the end of laparoscopic colorectal surgery would reduce the incidence of post operative pain, time spent in recovery room, improve patient's satisfaction, and reduce hospitalisation time

DETAILED DESCRIPTION:
Visits:

* The patient will arrive in the department the day before the surgical intervention (Day-1). During this preoperative visit (Day-1), the investigator

  * will preselect potentially eligible patients
  * will offer to participate to this study
  * will give the notice form to the patients
  * will present the research: objectives, benefits and constraints for the patients
* The intervention day (Day 0):

The investigator will collect the signed consent form after having ascertained the understanding of the notice form by the patient and checking the inclusion and non-inclusion criteria.

The randomization will be done via the eCRF module (allocation group and number) and the preoperative data registration in the eCRF.

Surgical Intervention (Day 1):

All patients will receive standard anaesthesia using sufentanyl, propopol, cisatracurium and sevoflurane. Prevention of nausea and vomiting is performing using Apfel score. Anti microbial prophylaxis is performed according recommendations.

All patients will receive post operative multimodal analgesia using intravenous lidocaine, acetaminophene, ketaminophene, and morphine if NRS (numerating rating scale) > 3 At the end of the surgery, patients in the experimental group will receive a bilateral ultrasound guided quadratus lumborum block with 15 ml of 3,75 mg/mg of ropivacaine. Patients in the control group will not receive the block

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients operated of a scheduled laparoscopic colorectal surgery
* Patients having given consent in the mannen described in Article L1122-1-1 of the Public Health Code
* Patients affiliated with asocial security regimen or beneficiary of such a regimen

Exclusion Criteria:

* Renal insufficiency (ie glomerular filtration output < 35 ml/min)
* Patients with chronic inflammatory bowel disease
* Body mass index > 35 kg/m2
* Chronic pain with opiates
* Patients with cognitive troubles
* Coagulation disorders (platelets count < 80G/L, PT< 50%, V factor < 50%)
* Pregnancy
* Breastfeeding
* Local anesthesics (amide class) allergy
* Laparotomy conversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Morphine Consumption in milligramme | 8 AM (ante meridiem) the day after surgery
  Once the patient is transferred in post operative surgical service, assessment of the primary outcome will be done by the nurse in charge of the patient

SECONDARY OUTCOMES:
NRS (Numeric rating scale) | At the entrance of recovery room, at day 1 and Day 2 after surgery
  Numerating rating score evaluating pain and variating from 0 (No pain) to 10 (Maximum Pain), done by nurses in operating room and in post operative surgical service
Post Operative recovery: QUO-R4O questionnaire | At Day 1 and day 15 after surgery
  Quo 40 score is a postoperative recovery score above 200 points (40 is worst score and 200 the best score) validated by Myles et al in 2001.
Time spent in recovery room (in minutes) | At the output of recovery room ie until 6 hours after intervention
  Assessment of time spent in recovery room (ie: entrance in recovery room until Aldrede score is >9) performed by nurses

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vignaud, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France